CLINICAL TRIAL: NCT00959478
Title: Emergency Department Brief Intervention to Increase Carbon Monoxide Detector Use
Acronym: ProjectCODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lara McKenzie (Other)
Responsible Party: Sponsor-Investigator, Lara McKenzie, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HD057155; Grant No.: R01HD057155
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Intervention-carbon Monoxide Alarm + Educational Tool; Control- Usual Care Flyer on Carbon Monoxide
Keywords: Carbon Monoxide (CO); Carbon Monoxide Poisoning; Carbon Monoxide Alarm/Detector; Precaution Adoption Process Model (PAPM); Injury Prevention; Emergency Department
MeSH Terms: conditions — Carbon Monoxide Poisoning; Emergencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Educational tool & Carbon Monoxide Alarm (Experimental): Parents will be randomly assigned into a control and intervention group. Both groups will complete a computer based survey at enrollment and at their home visits occuring two weeks and approximately six months following enrollment. Participants will be given the following materials at enrollment.
  Intervention:
  * Fast Facts about Carbon Monoxide Educational Tool
  * Kidde Nighthawk Carbon Monoxide Alarm
  Control:
  - Central Ohio Poison Control Center Flyer
  Interventions: Behavioral: Educational Tool & Carbon Monoxide Alarm

INTERVENTIONS:
Behavioral: Educational Tool & Carbon Monoxide Alarm — Based on the recommendations from the expert panel and focus group meetings, Fast Facts about Carbon Monoxide was developed to be an educational tool aimed at helping parents understand the dangers of CO and the need CO alarms in every home. In addition, this tool will help parents select and purchase the correct CO alarm, as well as properly install and maintain the alarm in their home. Each parent assigned to the intervention group will be given a Fast Facts about Carbon Monoxide educational tool and a Kidde Nighthawk Carbon Monoxide Alarm at enrollment.
  Other Names: Fast Facts about Carbon Monoxide Educational Tool

SUMMARY:
Carbon Monoxide (CO) exposure kills and injures thousands of children and families each year. Although there is growing concern about the need to increase carbon monoxide detector use, little is known about how best to do so, especially for low-income families. The objective of this research is to determine whether a brief intervention, Project Carbon Monoxide Detector Education (Project CODE), will increase CO detector use. For this study, parents of children, 18 years or younger, will be randomly assigned to receive Project CODE (an educational tool and a CO detector) or usual care (a flyer on CO poisoning); both of which will be delivered in the Pediatric Emergency Department (PED) examination rooms. The use of a CO detector and the participant's current stage in the theory of stage-based behavior change-the Precaution Adoption Process Model (PAPM), will be assessed at enrollment and then again at the home visits which will occur two-weeks and six-months following the PED visit. The investigators hypothesize that parents receiving Project CODE will have working CO detectors and will be further along in the PAPM than parents in the control group at the two-week and six-month home visits. The long term goal of this research is to reduce the number of injuries and deaths from CO poisoning.

DETAILED DESCRIPTION:
Poisoning from Carbon Monoxide (CO) is among the leading causes of non-fatal injuries treated in US hospital emergency departments and accounts for approximately 500 unintentional deaths each year. Known effective countermeasures to detect CO and reduce CO poisoning exist, yet are not routinely utilized. Although there is increasing concern about the need to increase CO detector use, little is known about how best to do so, especially for low income families. This research aims to address this gap, by applying a theory of stage-based behavior change-the Precaution Adoption Process Model PAPM)-to a brief intervention feasible for a busy emergency department setting. A randomized trial will be conducted involving 300 families with children 18 years or younger. In the Pediatric Emergency Department (PED), eligible parents will randomly be assigned to receive the Project CODE intervention (an educational tool and a CO detector) or usual care (a flyer on CO poisoning). The use of a CO detector and participant's PAPM stage will be assessed at enrollment and again at follow-up home visits occurring two-weeks and six-months following the PED visit. We hypothesize that parents receiving Project CODE will have working CO detectors and will be further along in the PAPM than parents in the control group at a two-week and six-month follow-up home visits. By examining the extent to which the intervention increases CO detector use, these findings will also demonstrate how innovative health communications (brief interventions delivered in the PED) can reduce the risk of injuries among vulnerable children. This research builds on and extends the investigators' previous work on behavioral theory, injury prevention interventions delivered in the PED, and development and evaluation of interactive educational tools for safety practices. The specific aims of this project are as follows: Aim 1-Determine whether a brief intervention will increase CO detector use and PAPM stage among parents whose children are being seen in a PED compared to parents of children receiving routine care CO flyer; and Aim 2-Determine whether and to what extent socioeconomic status moderates the effect of the intervention. Findings from this research study will have both theoretical and practical applications for improving injury prevention services in PEDs. This single-site efficacy trial is the first step in determining whether a brief intervention in the PED will successfully increase CO detector use.

ELIGIBILITY:
Inclusion Criteria:

* Age: The child being treated in the PED must be 18 years old or younger. The parent/guardian of the child being treated must be at least 18 years of age.
* Current/Previous Enrollment: The participant must only enroll in the study once. A participant may not re-enroll in the study after completing any step of the study nor can they enroll as a result of an additional trip to the PED with the same child or a sibling of that child.
* English speaking: Participants must feel comfortable answering survey questions that are written in English to be eligible for Project CODE.
* Parent/Guardian: The parent/guardian is the actual study participant, not the child, even if the child is eighteen years-old. The child treated in the PED must be accompanied by an English-speaking adult and that adult must be the person responsible for ensuring the child's safety in his/her home. The child must live with the adult most of the time.
* Reason for PED visit: Information regarding the nature of the child's visit will be obtained by reviewing PED triage information via EPIC and must be for an injury or a medical complaint.
* Place of Residence: Study participants must live in Franklin County (Columbus, Ohio and surrounding area).

Exclusion Criteria:

* Children being seen for possible sexual or physical abuse, neglect, behavioral problems, self inflicted harm or a suicide attempt.
* Children that must see a doctor immediately or are presenting with a critical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Observation of working carbon monoxide alarms | Two-weeks and six-months following enrollment

SECONDARY OUTCOMES:
Behavioral profile and Precaution Adoption Process Model(PAPM)stage | Two-weeks and six-months following enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lara B. McKenzie, PhD, Principal Investigator — Center for Inury Research and Policy, The Research Institute at Nationwide Children's Hospital
Locations (1):
- The Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] McKenzie LB, Roberts KJ, Kaercher RM, Collins CL, Comstock RD, Fernandez S, Abdel-Rasoul M, Casavant MJ, Mihalov L. Paediatric emergency department-based carbon monoxide detector intervention: a randomised trial. Inj Prev. 2017 Oct;23(5):314-320. doi: 10.1136/injuryprev-2016-042039. Epub 2016 Dec 22. PMID 28007971
- See also: The Center for Injury Research and Policy, The Research Institute at Nationwide Children's Hospital — http://www.injurycenter.org